CLINICAL TRIAL: NCT02150772
Title: Shear Wave Elastography in the Diagnosis and Risk-stratification of Thyroid Nodules - a Prospective Study
Brief Title: The Diagnostic Value of Shear Wave Elastography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Kristine Zøylner Rubeck, MD, University of Aarhus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SWE-diag 042014
Record Dates: First submitted 2014-04-14; First posted 2014-05-30 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

ARMS (1):
- Shear Wave Elastography (Other): All included patients have SWE performed
  Interventions: Procedure: Shear Wave Elastography (SWE)

INTERVENTIONS:
Procedure: Shear Wave Elastography (SWE)

SUMMARY:
Background: The main goal when diagnosing thyroid nodules, is to differentiate the few malignant from the overwhelming background of benign nodules. Currently available pre-operative tests are unable to rule out malignancy in a subset of patients and diagnostic thyroid surgery is necessary. Therefore, there is a need to develope the diagnostic tools for pre-operative diagnostic work-up of thyroid nodules.

The study will investigate a novel ultrasonographic technique called Shear Wave Elastography (SWE) in the pre-operative evaluation of thyroid nodules.

Aim:

To evaluate the diagnostic value of SWE in the pre-operative diagnosis of thyroid nodules in a tertiary surgical center.

Perspectives:

An optimization of the pre-operative risk-stratification and diagnosis of thyroid nodules can reduce unnecessary thyroid surgery, with a reduction in morbidity and better use of the economic and surgical resources.

ELIGIBILITY:
Inclusion Criteria:

* Nodules in the thyroid size more than 1 cm and patient undergoing thyroid surgery

Exclusion Criteria:

* Not undergoing thyroid surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Elasticity Index | same day
  Elasticity Index is obtained by SWE.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Z Rubeck, MD, Principal Investigator — Dep. of otorhinolaryngology, Aarhus University Hoapital; Viveque E Nielsen, MD PhD, Study Director — Dep. of oto-rhinolarymgology and Head and Neck surgery, Aarhus Universtity Hospital; Steen J Bonnema, PhD, DMSc, Study Chair — Dep. of Endocrinology, Odense University Hospital; Marie Louise Jespersen, MD, Study Chair — Dep. of Pathology, Aarhus University Hospital; Peer Christiansen, DMSc, Study Chair — Dep. og General Surgery, Aarhus University Hospital
Locations (1):
- Øre-Næse-Halsafdeling H, Aarhus University Hospital, Aarhus C, Denmark

REFERENCES:
- [Derived] Bakkegaard P, Londero SC, Bonnema SJ, Nielsen VE, Jespersen ML, Swan KZ. Risk-stratification of thyroid nodules examined by 18FDG-PET/CT while ensuring congruity between imaging and histopathological localization. Eur Arch Otorhinolaryngol. 2021 Dec;278(12):4979-4985. doi: 10.1007/s00405-021-06733-5. Epub 2021 Mar 13. PMID 33713190